CLINICAL TRIAL: NCT00657566
Title: SIS Multicenter Study of Duration of Antibiotics for Intraabdominal Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Robert Sawyer, MD, PI, National Institute of General Medical Sciences (NIGMS)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13447; 1R01GM081510-01 (NIH)
Record Dates: First submitted 2008-04-10; First posted 2008-04-14 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Peritonitis
Keywords: intraabdominal; peritonitis; sepsis; duration; antibiotics
MeSH Terms: conditions — Peritonitis; Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): antibiotics received for up to two days following normalization of white blood cell count, temperature, and gastrointestinal function
  Interventions: Other: duration of antibiotics
- 2 (Experimental): 4 +/- 1 days of antibiotics
  Interventions: Other: duration of antibiotics

INTERVENTIONS:
Other: duration of antibiotics — 4 +/- 1 days of antibiotics
  Other Names: short course
  Arms: 2
Other: duration of antibiotics — active comparator antibiotics given until 2 days after resolution of fever, elevated white blood cell count, and gastrointestinal dysfunction.
  Other Names: long course
  Arms: 1

SUMMARY:
The major hypothesis to be tested is that the treatment of intraabdominal infections that have been adequately treated operatively or by percutaneous techniques with three to five days of antibiotics will result in outcomes equivalent to the current standard where treatment is carried out until the patient has returned to normal (normal white blood cell count, temperature, and intestinal function), and that patients treated for three to five days will receive fewer days of antibiotics than the control group that has traditionally received seven to 14 days of treatment.

DETAILED DESCRIPTION:
Overall, this is a prospective, randomized, single-blinded (analysis), fifteen-center study using intent to treat analysis. Patients will be identified and after informed consent is obtained, will be randomized to receive antibiotics for 3 to 5 days (4 ± 1 days) after the initial surgical or percutaneous intervention or antibiotics until two calendar days after the patient's white blood cell count, systemic temperature, and gastrointestinal function have normalized (maximum of 10 days). The primary endpoint is the composite rate of in-hospital death and/or recurrence of intraabdominal infection and/or occurrence of surgical site (wound) infection. Secondary endpoints include the occurrence of any infection at any site and infection with antibiotic-resistant pathogens. Patient data through the thirty days following the initial intervention or until hospital discharge (whichever is longer) will be tracked

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 16 at some sites,(≥ 18 at UVA)
* ability to obtain informed consent from the subject or surrogate
* Presence of an intraabdominal infection requiring any duration of hospitalization and managed with open, laparoscopic, or percutaneous intervention.
* A peripheral white blood cell count of > 11,000/mm and/or temperature ≥ 38.0 C with in 24 hours or gastrointestinal dysfunction sufficient to prevent intake of normal diet within 24hrs of initial operative or percutaneous intervention.
* Adequate source control in the opinion of the local investigator and PI. Source control is defined as any procedure that stops the ongoing contamination of the peritoneal cavity and removes the majority of the contaminated intraperitoneal contents to the extent that no further acute interventions are felt to be necessary.

Exclusion Criteria:

* age < 16 years at some sites(< 18 at UVA)
* Inability to obtain consent from the patient, parents, or surrogate
* Lack of adequate source control in the opinion of the local investigator or overall PI ( Robert Sawyer)
* High likelihood of death within 72 hours of initial intervention in the opinion of the local investigator or principal investigator
* Lack of any clinical improvement within 72 hours of initial intervention in the opinion of the local investigator or principal investigator.
* Planned relaparotomy
* Perforated gastric ulcer or duodenal ulcer treated within 24hours of the onset of symptoms
* Traumatic injury to the bowel (including iatrogenic or intra-operative) treated within 12 hours of injury
* Non-perforated, non-gangrenous appendicitis or cholecystitis
* Gangrenous appendicitis or peritonitis without confirmatory cultures or with cultures without bacterial or fungal growth
* Ischemic or necrotic intestine without perforation and without positive bacterial or fungal cultures
* Intraabdominal infection associated with active necrotizing pancreatitis
* Primary (spontaneous) bacterial peritonitis
* Intraabdominal infection associated with an indwelling continuous ambulatory peritoneal dialysis catheter.
* Primary skin closure of an open surgical incision in the presence of diffuse, non-localized peritonitis. Laparoscopic port sites ≥ 2cm may be closed
* Pregnancy
* Prior enrollment in this study
* Enrollment in another therapeutic trial

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2008-09; Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be percentage failure conditioned by assigned duration of antibiotic therapy (intent to treat analysis). | 30 days

SECONDARY OUTCOMES:
Failure rate for clinically evaluable patients receiving the appropriate duration of antibiotics | 30 days
failure rate for microbiologically evaluable patients | 30 days
rate of need for reintervention in the abdomen | 30 days
rate of surgical site infection | 30 days
rate of death within 30 days | 30 days
duration of hospitalization | 30 days
rate of intraabdominal or surgical site failure due to antimicrobial-resistant pathogens | 30 days
rate of any subsequent infection at a site other than the abdomen or the surgical site | 30 days
rate of infection at a non-abdominal, non-surgical site with a resistant organism | 30 days
rate of Clostridium difficile infection | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Sawyer, MD, Principal Investigator — University of Virginia
Locations (23):
- United States (22):
  - Maricopa Medical Center-Phoenix, Phoenix, Arizona
  - University of California Davis, Sacramento, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Univestity of Kansas, Kansas City, Kansas
  - Louisville-VA, Louisville, Kentucky
  - Louisville-University Hospital, Louisville, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Brigham and Womens, Boston, Massachusetts
  - Univeristy of Michigan, Ann Arbor, Michigan
  - Washington Universtiy, St Louis, Missouri
  - Wake Forest University, Winston-Salem, North Carolina
  - Case Western, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Pittsburgh VA, Pittsburgh, Pennsylvania
  - University of South Carolina, Columbia, South Carolina
  - Universtiy of Texas San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Virginia-Virginia Commonwealth University Hospital, Richmond, Virginia
  - University of Washington-Harborview, Seattle, Washington
  - University of Washington - University Hospital, Seattle, Washington
- St Michael's, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hedrick TL, Evans HL, Smith RL, McElearney ST, Schulman AS, Chong TW, Pruett TL, Sawyer RG. Can we define the ideal duration of antibiotic therapy? Surg Infect (Larchmt). 2006 Oct;7(5):419-32. doi: 10.1089/sur.2006.7.419. PMID 17083308
- [Derived] Sawyer RG, Claridge JA, Nathens AB, Rotstein OD, Duane TM, Evans HL, Cook CH, O'Neill PJ, Mazuski JE, Askari R, Wilson MA, Napolitano LM, Namias N, Miller PR, Dellinger EP, Watson CM, Coimbra R, Dent DL, Lowry SF, Cocanour CS, West MA, Banton KL, Cheadle WG, Lipsett PA, Guidry CA, Popovsky K; STOP-IT Trial Investigators. Trial of short-course antimicrobial therapy for intraabdominal infection. N Engl J Med. 2015 May 21;372(21):1996-2005. doi: 10.1056/NEJMoa1411162. PMID 25992746